CLINICAL TRIAL: NCT03510949
Title: The Use of Nasopharyngeal Airway as an Alternative to Laryngeal Mask Airway to Maintain Anaesthesia in Patients Undergoing Four-Lids Blepharoplasty
Brief Title: Nasopharyngeal Versus Laryngeal Mask Airway in Anaesthesia for Bilateral Blepharoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hala Salah El-Din El-Ozairy (Other)
Responsible Party: Sponsor-Investigator, Hala Salah El-Din El-Ozairy, Lecturer of Anaesthesia, ICU and Pain management, Faculty of Medicine, Ain Shams University, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R 48/2017
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Injury Throat
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Group N: Patients' nasal mucosa will be anaesthetized and vasoconstricted. The NPA will then be advanced into the dominant nostril along the septum horizontally.
  Group L: K-Y gel will be applied to the tip of the laryngeal mask (LMA) of appropriate size. The LMA will be introduced along the hard palate towards the hypopharynx until resistance is felt.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Other): Patients' nasal mucosa will be anaesthetized and vasoconstricted. K-Y gel will be applied to the tip of nasopharyngeal airway (NPA) of appropriate size. The NPA will then be advanced into the dominant nostril along the septum horizontally.
  Interventions: Device: Nasopharyngeal airway or laryngeal mask airway
- Group L (Other): K-Y gel will be applied to the tip of the laryngeal mask (LMA) of appropriate size. The LMA will be introduced along the hard palate towards the hypopharynx until resistance is felt.
  Interventions: Device: Nasopharyngeal airway or laryngeal mask airway

INTERVENTIONS:
Device: Nasopharyngeal airway or laryngeal mask airway — Comparing the incidence of postoperative soar throat with the use of nasopharyngeal airway versus laryngeal mask airway

SUMMARY:
General anaesthesia demands securing patient's airway either with endotracheal tube or laryngeal mask (LMA); however, both carry the disadvantage of postoperative soar throat. Nasopharyngeal airway (NPA) can be an alternative without the risk of postoperative soar throat.6 The primary end point of our study is to assess the incidence of soar throat with the use of NPA compared to LMA in patients receiving general anaesthesia during blepharoplasty.

DETAILED DESCRIPTION:
After approval of medical ethical committee at Ain-Shams University and obtaining written informed consent, 148 adult ASA II-III patients aged between 40 and 60 years old admitted to Ain-Shams university hospitals for blepharoplasty will be enrolled in this study.

Patients will then be randomly and evenly divided into two equal groups (74 patients each) using computer-generated list:

Group N: Patients' nasal mucosa will be anaesthetized and vasoconstricted. K-Y gel will be applied to the tip of nasopharyngeal airway (NPA) of appropriate size. The NPA will then be advanced into the dominant nostril along the septum horizontally.

Group L: K-Y gel will be applied to the tip of the laryngeal mask (LMA) of appropriate size. The LMA will be introduced along the hard palate towards the hypopharynx until resistance is felt.

Anaesthesia will be maintained by sevoflurane 3-4% and propofol infusion 0.5-1 mg.kg-1.hr-1.All patients will receive local infiltration anaesthesia given by the surgeon.

At the conclusion of surgery, sevoflurane and propofol infusion will be discontinued and patients will inhale 100% O2 till spontaneous recovery.

Recovery time will be recorded (defined as the time from discontinuation of anaesthetic drugs till response to verbal command).

Incidence of postoperative soar throat, unsteadiness, nausea and vomiting will be recorded as well as patient and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* consented patients, age: 40-60 years old, ASA II-III

Exclusion Criteria:

1. Uncontrolled hypertension (systolic blood pressure > 160 mmHg) or ischaemic heart disease.
2. Pre-existing coagulation defects or anticoagulation medication.
3. Renal impairment.
4. Recent upper respiratory tract infections, asthma, chronic obstructive pulmonary disease, and smoking.
5. History of obstructive sleep apnea.
6. Chronic drug or alcohol abuse.
7. Morbid obesity; BMI >40 or BMI >35 and experiencing obesity-related health conditions, such as high blood pressure or diabetes.
8. Allergy to any of the drugs used in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative soar throat | 2-4 hours postoperative
  presence or abscence of soar throat

CONTACTS AND LOCATIONS:
Overall Officials: Hala S El-Ozairy, MD, Principal Investigator — Anaesthesia department, faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided